CLINICAL TRIAL: NCT00276263
Title: Sarcosine (N-methylglycine) Trial for Individuals At Risk for Developing Schizophrenia and Related Disorders
Brief Title: Sarcosine Preventive Therapy for Individuals At High Risk for Schizophrenia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of participants
Sponsor: Herzog Hospital (Other)
Responsible Party: Principal Investigator, Heresco-Levi Uriel, Uriel Heresco-Levy, Herzog Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Heresco 3 CTIL; 101-06
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenias; Psychoses; Psychotic Disorders; Schizophrenic Disorders
Keywords: Schizophrenia prodrome; Sarcosine; Psychosis; NMDA receptor; Prevention
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Sarcosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sarcosine (N-methylglycine)

INTERVENTIONS:
Drug: Sarcosine (N-methylglycine) — Randomization to two treatment groups. One group treated with sarcosine 2 g/day for 16 weeks, the other group treated with placebo 2 g/day for 16 weeks.

SUMMARY:
The purpose of this study is to determine whether preventative treatment with sarcosine can reduce symptoms and delay/avoid disease progression in individuals defined as being in a prodromal stage of schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a neurodevelopmental disorder that affects approximately 1% of the general population and continues to be one of the major challenges of modern medicine due to the tremendous human suffering and economic costs that it involves. Once the diagnosis of schizophrenia or a related chronic psychosis has been made, the majority of patients will only partially respond to presently available pharmacological treatments and will be afflicted by long-standing deficits affecting all aspects of mental functioning.

This unfavourable outcome highlights the importance of preventive treatment for schizophrenia and related psychoses. The notion of early pharmacological intervention during the prodromal phase of these disorders has a dual aim: 1) to treat active prodromal symptoms and 2) to prevent further deterioration and progression toward the full-blown disorder and chronicity. Overall, it raises the possibility of preventing, delaying or ameliorating the onset of the diagnosable disorder. This type of intervention, although already in use in other medical branches and potentially ground-breaking for mental health delivery systems, has not been systematically assessed in the past. Recently, the development of improved criteria for detecting individuals at high risk for developing schizophrenia and related psychoses, has led to the first clinical trials that assessed the role of atypical antipsychotics (i.e., risperidone and olanzapine) for these subjects. The results of these studies indicate that significant clinical benefits nay be derived from early intervention but also point to the drawbacks of exposing patients at a very early stage of illness to antipsychotic drugs that are associated with debilitating (i.e. motor, metabolic) side effects.

The overall aim of the proposed project is to assess the efficacy and safety of the N-methyl-D-aspartate glutamate receptor (NMDAR) modulator, glycine transport inhibitor sarcosine (N-methylglycine) for the treatment of individuals fulfilling schizophrenia prodromal syndromes criteria. NMDAR's dysfunction plays a cardinal role in schizophrenia pathophysiology and the establishment of neurodevelopmental deficits. During the last decade it was demonstrated that pharmacological treatment with compounds that enhance NMDAR-mediated neurotransmission due to their agonistic activity at the NMDAR-associated glycine site (e.g. glycine, D-serine) leads to significant symptom reductions in chronic schizophrenia patients. Furthermore, preliminary findings suggest that glycine treatment may also be beneficial for patients at high risk for developing schizophrenia. By increasing glycine synaptic levels, sarcosine may generate improved therapeutic effects in high risk individuals. Sarcosine is a natural amino acid that has already been shown to reduce positive, negative and cognitive symptomatology in chronic as well as acute schizophrenia patients. Advantages of sarcosine vs. glycine site agonists use include the relatively low dose required and the lack of known side effects. Synthetic compounds conceptually similar to sarcosine are presently in various stages of development by major pharmacological companies.

In the proposed project, during a three-year period, 60 individuals fulfilling prodromal criteria will be randomly entered in a 16 week parallel group, double-blind, placebo controlled trial with 2 gr/day sarcosine, with an optional 8 week open-label extension. Clinical, neurocognitive, electrophysiological, amino acids (i.e. glycine, serine, glutamate) levels and genetic assessments will be performed during the study. The specific aims of the proposed project are: 1) to assess the efficacy and safety of sarcosine as active treatment for prodromal symptoms, 2) to assess sarcosine effects in terms of relevant amino acids serum levels, neurocognitive performance and relevant brain electrophysiological parameters and 3) to supply preliminary data in regard to the capacity of sarcosine treatment to delay/prevent conversion to full blown psychotic disorder. The overall importance of the proposed project consists of its potential to lay the foundations for an innovative type of treatment for schizophrenia prodromal states.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-seeking male or female outpatients, 12-45 years old
* Meet the definition of one or more prodromal syndromes according to the Criteria of Prodromal Syndromes (COPS) derived using the SIPS/SOPS scales.
* Possession of a level of understanding sufficient to communicate with the investigator and to understand the nature of the study
* Agreement to participate in the study and sign informed consent. Minors will be required to give written informed consent with written consent from a parent or guardian

Exclusion Criteria:

* Meeting criteria for past or current DSM-IV psychotic disorder
* Judged clinically to suffer from a psychiatric disorder (e.g. ADHD, mania, depression) that could account for the inclusion symptoms
* Judged clinically to be at suicidal or homicidal risk
* Symptoms judged clinically to be sequelae of drug or alcohol abuse
* IQ of less than 80
* Seizure disorder without a clear or resolved etiology
* Female patients who are pregnant or lactating; female patients who are not pregnant or lactating, if sexually active, must be using medically accepted means of contraception
* Taking non-protocol psychiatric medications within two weeks of randomization or depot psychiatric medications three months prior to study entry
* Individuals suffering from an unstable and/or untreated medical disorder will not be entered in the study

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Study Completion 2009-06

PRIMARY OUTCOMES:
Sarcosine vs. placebo in subjects at risk for developing schizophrenia:efficacy and safety. | 16 weeks
Sarcosine is superior to placebo in the treatment of positive, negative, and cognitive (disorganized) symptoms. Safety assessed with UKU scale, vital signs measurements and laboratory parameters (SMA-20, CBC, UA) | 16 weeks
Sarcosine vs. placebo in the treatment of neurocognitive dysfunction | 16 weeks

SECONDARY OUTCOMES:
To assess the efficacy of sarcosine in delay/prevention of illness progression. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Heresco-Levy, M.D., Principal Investigator — Ezrath Nashim - Herzog Hospital / Hadassah Medical School; Bernard Lerer, M.D., Principal Investigator — Department of Psychiatry, Hadassah Hospital
Locations (2):
- Israel (2):
  - Ezrath Nashim - Herzog Memorial Hospital, Jerusalem
  - Department of Psychiatry, Hadassah Hospital and Community Clinics, Jerusalem